CLINICAL TRIAL: NCT02444078
Title: Effects of a Long-term Exercise Program on Functional Ability in People With Dementia Living in Nursing Homes: a Cluster Randomised Controlled Trial. The LEDEN Study
Brief Title: Effects of Exercise on Functional Ability in People With Dementia in Nursing Homes:a Cluster Randomised Controlled Trial
Acronym: LEDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/14/7292; 2014-A01713-44 (Other: ID-RCB)
Record Dates: First submitted 2015-04-24; First posted 2015-05-14 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer Disease; Dementia; Physical activity; Functional ability; Disability; Functional limitation
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Exercise sessions will be done in groups of three-to-eight persons; whilst being a group-based exercise program, participants will be guided and the exercises will be adapted in an individual basis, which may increase adherence and compliance rates.
  Interventions: Other: Exercise
- Social activity (Active Comparator): Participants in this group will participate in group-based activities such as music (percussion instruments), arts and board games; no intervention on physical activity will be provided to these participants.
  Interventions: Other: Social Activity

INTERVENTIONS:
Other: Exercise — Exercise training will take place in the NH, twice weekly, around 60 minutes per session (session duration can be shorter during the first weeks of intervention according with participants' physical capacity), during 6 months; interval between two exercise sessions will be of at least 48 hours. The exercise program will be a multicomponent training, with exercises specifically developed to improve participants' flexibility (10 minutes), coordination and balance (10 minutes), muscle toning (10 minutes), and cardiorespiratory capacity (25 minutes). The exercise intensity targeted will be moderate. All exercise sessions will be accompanied by music.
  Arms: Exercise
Other: Social Activity — Interventionists will be health professionals external to the NH, preferentially psychologists. Interventions will take place in the NHs, at the same frequency and duration than the exercise intervention (twice weekly, 60 minutes per session, during 6 months).
  Arms: Social activity

SUMMARY:
This is a cluster randomised controlled trial composed of two research arms: exercise training group (experimental group) and a social activity group (control group).

DETAILED DESCRIPTION:
The recruitment process will be made only in NHs (Nursing Home) where the staff will have voluntarily accepted to participate in the study. We estimated to recruit 140 PWD (person with dementia) from around six-to-eight NHs (i.e., in average a minimum of 18 and a maximum of 24 PWD per NH). NHs constitute the unit of randomisation; NHs will be randomised to study groups using a 1:1 ratio (it means that all the participants living in a particular NH will participate in either the exercise training or the social activity). The randomisation will be stratified by the prevalence of dementia among NH residents; this stratification will provide homogeneity across research's arms, increasing thus the comparability among groups and producing then reliable results. Randomisation will be done by a statistician not involved in the LEDEN study. Allocation concealment will be ensured by the use opaque sealed envelopes. The randomisation list will be kept in a electronic, password-locked file matching the name of participants to their research identification number and their group allocation. Given the nature of the LEDEN intervention (exercise training, i.e., a behavioural intervention) and since the main outcome measure, i.e., participants' ability in executing ADLs, of the the study requires that the outcome assessor knows how participants cope in their daily life, LEDEN is a unblinded study

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Alzheimer's disease, vascular or mixed dementia according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV);
* MMSE ≤ 20 (out of 30);
* living in one of the participating NHs for at least 3 months at the moment of baseline measurements (this time period will allow NH staff to have a good knowledge about the patient and about recent changes in his/her health status);
* to be able of walking at least 4 meters (with walking devices if needed but without human assistance);
* to be able to rise from a chair without help or with minimal human assistance.

Exclusion Criteria:

* Mild dementia, illustrated by a MMSE > 20 (out of 30)
* Terminal illness with life expectancy less than 6 months;
* Diagnosis of Parkinson's disease;
* Diagnosis of dementia with Lewy bodies;
* Unstable cardiovascular condition or any other health condition that might be deteriorated by physical exercise;
* Planned transfer from the NH to another NH/home or to surgery during the 6-month period of intervention;
* Already participating in physical exercise ≥ 2 times/week in the last 2 months prior to the date of baseline assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Functional ability | 6th month
  (ADL performance) as assessed by the Alzheimer Disease Cooperative Study (ADCS) ADL-sev. This is a 19-item scale measuring the ability to perform basic (e.g., bathing, toileting) and instrumental (e.g., turning faucet/lights on/off) ADLs in the last four weeks. The ADCS-ADL-sev was specifically validated for people with moderate or severe Alzheimer's disease (AD), i.e., the large majority of PWD in NHs. Scores in this scale vary from 0 to 54, with higher scores indicating better functional ability.

SECONDARY OUTCOMES:
Change of Functional ability | Change and evolution at different time points: baseline, 3-month intervention, Post-intervention (6month), 3-month follow-up (9 month), 6-month follow-up (12 month)
  ADL performance) as assessed by the Alzheimer Disease Cooperative Study (ADCS) ADL-sev. This is a 19-item scale measuring the ability to perform basic (e.g., bathing, toileting) and instrumental (e.g., turning faucet/lights on/off) ADLs in the last four weeks. The ADCS-ADL-sev was specifically validated for people with moderate or severe Alzheimer's disease (AD), i.e., the large majority of PWD in NHs. Scores in this scale vary from 0 to 54, with higher scores indicating better functional ability.
Physical function | Baseline, Post-intervention (6 month)
  as assessed by the Short Physical Performance Battery (SPPB) (score from 0 to 12).
Cost-effectiveness of the interventions | 12 month (end of study)
Falls and fractures | 12 month (end of study)
Cognitive function | Baseline, Post-intervention (6month)
  as assessed by the Mini-Mental State Examination (MMSE).
Behavioural and psychological symptoms of dementia (BPSD) | Baseline, Post-intervention (6 month)
  as assessed by the Neuropsychiatric Inventory - Nursing Home version (NPI-NH).
Pain | Baseline, Post-intervention (6 month)
  as assessed by the Algoplus scale
Nutritional status | Baseline, Post-intervention (6 month)
  as assessed by the Mini Nutritional Assessment (MNA).

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROLLAND, MD, Principal Investigator — Toulouse University Hospital (CHU Toulouse)
Locations (8):
- France (8):
  - Résidence d'Automne de Bruay sur Escaut, Bruay-sur-l'Escaut
  - Korian Le Castelli, L'Huisserie
  - Korian Pontlieue, Le Mans
  - Résidence Les Lauriers de Plaisance, Neuilly-Plaisance
  - Korian Croix Périgourd, Saint-Cyr-sur-Loire
  - Résidence d'Automne de Notre Dame de Sanhilac, Sanilhac
  - Résidence Les Jardins de Sermaize, Sermaize-les-Bains
  - Korian Vill'Alizé, Thise

REFERENCES:
- [Result] de Souto Barreto P, Cesari M, Denormandie P, Armaingaud D, Vellas B, Rolland Y. Exercise or Social Intervention for Nursing Home Residents with Dementia: A Pilot Randomized, Controlled Trial. J Am Geriatr Soc. 2017 Sep;65(9):E123-E129. doi: 10.1111/jgs.14947. Epub 2017 May 19. PMID 28542742
- [Result] de Souto Barreto P, Denormandie P, Lepage B, Armaingaud D, Rapp T, Chauvin P, Vellas B, Rolland Y. Effects of a long-term exercise programme on functional ability in people with dementia living in nursing homes: Research protocol of the LEDEN study, a cluster randomised controlled trial. Contemp Clin Trials. 2016 Mar;47:289-95. doi: 10.1016/j.cct.2016.02.004. Epub 2016 Feb 13. PMID 26883281